CLINICAL TRIAL: NCT02613091
Title: Effect of Clemastine Fumarate on Color Vision in Healthy Controls
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Ari Green, MD, MCR, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Clemastine Color Vision
Record Dates: First submitted 2015-10-23; First posted 2015-11-24 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Subjects
Keywords: volunteers
MeSH Terms: interventions — Clemastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clemastine (Experimental): This group will receive 8mg of clemastine daily.
  Interventions: Drug: Clemastine fumarate

INTERVENTIONS:
Drug: Clemastine fumarate — 4mg 2x day clemastine fumarate orally.

SUMMARY:
In a1972 study in the French Annals of Pharmaceuticals, Laroche and Laroche reported that the drug clemastine has a negative effect on patients' color discrimination, which is the ability to distinguish different hues and arrange them in the correct order. In an upcoming clinical trial studying the effect of clemastine on vision outcomes, our lab aims to assess color visual performance adding assessment of color defectiveness as a clinical endpoint. Color defectiveness is the ability to see certain colors, and is commonly referred to as color-blindness. Color discrimination and defectiveness can be related, but do not always correlate. This study aims to detect the effect, if any, that clemastine has on color defectiveness in healthy controls, which could confound its use as an outcome endpoint in future clinical trials relating to clemastine.

DETAILED DESCRIPTION:
Additional evaluation of pharmacokinetic data will be performed to confirm pharmacokinetic measures and correlate blood levels of drug to color performance if seen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy control

Exclusion Criteria:

* Preexisting ophthalmologic conditions such as optic neuritis, macular star, glaucoma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline cone contrast test score at 3 weeks | baseline, 3 day, 3 week
  Cone contrast and color vision testing to be performed at all 3 study visits

SECONDARY OUTCOMES:
Change from baseline Lanthany D15 score at 3 weeks | baseline, 3 day, 3 week
  Lanthany D15 test to be administered at all 3 study visits. Score determined by number of "crossings" as outlined in the following link http://www.richmondproducts.com/files/8113/1550/0538/FR_15_Farnsworth_and_LanthonyD15_Instructions_Rev_1.7_0506.pdf

CONTACTS AND LOCATIONS:
Overall Officials: Ari Green, MD, MCR, Principal Investigator — UC San Francisco
Locations (1):
- Sandler Neurosciences Building, Neurological Clinical Research Unit, San Francisco, California, United States

REFERENCES:
- [Background] Laroche. Modification of color vision elicited by the use of normal therapeutical dosage of some drugs. French Annals of Pharmaceuticals. 1972.